CLINICAL TRIAL: NCT06301399
Title: A Study on the Efficacy and Safety of Rituximab When Combined With Prior Targeted Therapy and Checkpoint Immunotherapy as Second-line or Later Therapy in Patients With Advanced Hepatocellular Carcinoma
Brief Title: Rituximab Combined With Prior Therapy in Advanced Hepatocellular Carcinoma: Efficacy & Safety Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Rituximab01
Record Dates: First submitted 2024-02-16; First posted 2024-03-08 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-02

CONDITIONS: Advanced Hepatocellular Carcinoma
Keywords: rituximab; Advanced Hepatocellular Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rituximab+PD-1 or PD-L1 inhibitors+targeted therapy (Experimental): Rituximab: Dissolve 375mg/m2 in 0.9% sodium chloride injection, dilute to a concentration of 1 mg/mL of rituximab, intravenous infusion every 3 weeks until tumor progression or intolerable toxic reactions occur. The recommended initial infusion rate is 50mg/h; After the initial 60 minutes, an increase of 50mg/h can be made every 30 minutes until the maximum speed is 400mg/h. The starting rate of rituximab infusion in the future can be 100mg/h, increasing by 100mg/h every 30 minutes until the maximum rate is 400mg/h.
  PD-1 (or PD-L1) inhibitors and targeted drugs: Select first-line PD-1 (or PD-L1) inhibitors and VEGFR targeted drugs according to clinical routine treatment, and administer according to the original first-line combination therapy dosage until progression or intolerable toxic reactions occur.
  Interventions: Drug: Rituximab+PD-1 or PD-L1 inhibitors+targeted therapy

INTERVENTIONS:
Drug: Rituximab+PD-1 or PD-L1 inhibitors+targeted therapy — Rituximab: Dissolve 375mg/m2 in 0.9% sodium chloride injection, dilute to a concentration of 1 mg/mL of rituximab, intravenous infusion every 3 weeks until tumor progression or intolerable toxic reactions occur. The recommended initial infusion rate is 50mg/h; After the initial 60 minutes, an increase of 50mg/h can be made every 30 minutes until the maximum speed is 400mg/h. The starting rate of rituximab infusion in the future can be 100mg/h, increasing by 100mg/h every 30 minutes until the maximum rate is 400mg/h.

SUMMARY:
Evaluation of the efficacy and safety of adding rituximab after failure of target immunotherapy in the Posterior treatment of advanced hepatocellular carcinoma

DETAILED DESCRIPTION:
Evaluation of the efficacy and safety of adding rituximab after failure of target immunotherapy in the Posterior treatment of advanced hepatocellular carcinoma

ELIGIBILITY:
Inclusion Criteria:

* 1)written informed consent signed prior to enrolment.
* 2) Age 17-79 years old (including boundary), male or female;
* 3) Subjects with histologically or cytologically confirmed advanced hepatocellular carcinoma (HCC), or clinical diagnosis that meets the American Association of Liver Diseases (AASLD) diagnostic criteria for hepatocellular carcinoma
* 4) Previous progression or intolerance after failure to target, immunization, or conventional therapy (including TKI, ICI, chemotherapy, VEGF monoclonal antibody, or ICI combined with TKI/VEGF monoclonal antibody/chemotherapy)
* 5) 2 weeks after the end of previous systemic therapy ≥ the first dose of this study, and the treatment-related AEs recovered to NCI-CTCAE ≤ Grade 1 (except for alopecia)
* 6) Child-Pugh liver function rating within 7 days prior to the first dose of the study drug: A grade and good B grade (≤ 7 points)
* 7) Phase B or C as assessed by BCLC or Phase III as assessed by CNLC
* 8) At least one measurable target lesion as assessed by the investigator according to the requirements of mRECIST v1.1 within 4 weeks prior to the first dose
* 9) Have adequate organ function (without receiving blood transfusion, erythropoietin, granulocyte colony-stimulating factor, albumin, or other medical support within 14 days prior to initiation of study drug therapy)
* 10) If the patient has HBsAg(+) or HBcAb(+), HBV-DNA must be < 2500 copies/mL or < 500 IU/mL or < upper limit of normal (ULN) to be enrolled, and those with elevated HBV-DNA must agree to receive nucleoside anti-hepatitis B virus therapy. Subjects who are negative for HCV antibody (-) or HCV-RNA are allowed to enroll, if HCV-RNA is positive, they need to agree to receive local standard standard antiviral therapy, and subjects must have ALT, AST, ≤ 3×ULN to enroll, and subjects with hepatitis B and C co-infection need to be excluded (HBV-DNA and HCV-RNA are positive)
* 11) Patients with cured hepatitis C are acceptable, and the lower limit of detection of HCV RNA < test center before starting study drug treatment
* 12) ECOG PS score: 0-1
* 13) Expected survival ≥ 12 weeks
* 14) Male or female of childbearing potential who are willing to use contraception in the trial, and females of childbearing potential must have a pregnancy test within 7 days prior to the first dose with a negative result
* 15)CD20 positive and CD20 scattered (non aggregated) distribution in tumors

Exclusion Criteria:

* 1) Known hepatocholangiocarcinoma, mixed cell carcinoma, or fibrolamellar cell carcinoma
* 2) History of hepatic encephalopathy within 6 months prior to the first dose of this study
* 3) Portal hypertension with endoscopic red signs, or those who are considered by the investigator to have a high risk of bleeding or who have had esophageal or gastric variceal bleeding within 6 months before the first dose
* 4) Symptomatic brain or meningeal metastases (unless the patient has been >treated for 3 months, there is no evidence of progression in imaging results within 4 weeks before the first dose, and tumor-related clinical symptoms are stable)
* 5) The patient has human immunodeficiency virus (HIV) or active tuberculosis, or other uncontrolled active infection
* 6) Those who have undergone major surgery within 4 weeks before enrollment, and those who have had bone marrow biopsy, open biopsy, and intracranial biopsy within 7 days before screening
* 7) Those who have other malignant tumors in the past 5 years and have not been effectively controlled, except for carcinoma in situ of the cervix, squamous cell carcinoma of the skin or localized basal cell skin cancer
* 8) Known history of severe allergy to any monoclonal antibody or study drug excipient
* 9) Pregnant or lactating women
* 10) Other reasons judged by the investigator to be unsuitable for participating in this study

Ages: 17 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | from the date of enrollment to death from any cause. (assessed up to 12 months）
  mRESIST

SECONDARY OUTCOMES:
PFS | from the date of enrollment to death from any cause. (assessed up to 12 months）
  mRESIST
OS | from the date of enrollment to death from any cause. (assessed up to 12 months）
  mRESIST
DoR | from the date of enrollment to death from any cause. (assessed up to 12 months）
  mRESIST
DCR | from the date of enrollment to death from any cause. (assessed up to 12 months）
  mRESIST

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality, China